CLINICAL TRIAL: NCT05873829
Title: The Effect of Hand-Foot Exercises on Platinum-Based Chemotheraphy Induced Peripheral Neuropathy Related Pain Severity, Falls and Quality of Life in Colorectal Cancer
Brief Title: Hand-Foot Exercises for Chemotheraphy Induced Peripheral Neuropathy Pain, Falls and Quality of Life in Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, İlayda EROĞLU, Research Assistant, Gulhane Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-50687469-929-1800
Record Dates: First submitted 2023-05-16; First posted 2023-05-24 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2023-05

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Colorectal Cancer
Keywords: Colorectal cancer, Peripheral Neuropathies,Nursing
MeSH Terms: conditions — Colorectal Neoplasms; Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: The patients, whose written and verbal consents were obtained in accordance with the inclusion criteria, were randomly assigned to the intervention and control groups.
  Hand-foot exercises were applied to the patients in the intervention group. The patients in the control group did not undergo any intervention other than standard care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Hand-foot exercises were applied to the intervention group.
  Interventions: Other: Hand-foot exercises
- Control Group (No Intervention): No intervention other than standard care was applied to the control group.

INTERVENTIONS:
Other: Hand-foot exercises — Hand-foot exercise program consists of 5 hand and 5 foot exercises, and a total of 15 minutes of simple hand-foot exercises. The exercise program is applied 3 times a day, 3 days a week. The tennis ball and the towel that used in the exercise program, the booklet which containing the exercise explanations and the video link showing the implementation of the exercises were provided by the researcher.
  Arms: Intervention Group

SUMMARY:
Colorectal cancer is the 4th most common cancer in the world among all cancer types. Chemotherapy-induced peripheral neuropathy is a common and serious side effect caused by chemotherapeutic agents, especially platinum analogues, taxanes, vinca alkaloids and bortezomib. The most commonly used chemotherapeutic agents in the treatment of colorectal cancers are platinum analogues It is known that oxaliplatin, one of the platinum analogues, causes 85-96% of chemotherapy-induced peripheral neuropathy. The most common symptoms of chemotherapy-induced peripheral neuropathy are; numbness, paresthesia, dysesthesia, pain, hypersensitivity to cold or heat, tingling, muscle cramps, distal weakness, gait disturbances, balance disorders, and impaired movement. Oxaliplatin, which is frequently used in the treatment of colorectal cancer, causes symptoms of both acute and chronic chemotherapy-induced peripheral neuropathy. There is no proven method in the treatment of chemotherapy-induced peripheral neuropathy. However, various pharmacological and non-pharmacological approaches are applied in its preventive and symptomatic treatment. Exercise and physical therapy interventions; It is stated that it improves strength, balance and other functional disorders in patients, reduces symptoms, and reduces the risk of falling by affecting gross motor dysfunctions such as balance and gait abnormalities. However, the limitations of studies on this subject in the literature draw attention. This situation suggests that new methods that can be applied in the care of cancer patients who develop peripheral neuropathy due to chemotherapy should be developed in the field of nursing. This research is the first study to evaluate the effect of hand-foot exercises on colorectal cancer patients who developed peripheral neuropathy due to platinum-based therapy. Research results; Alleviation of KBPN-induced pain and prevention of falls are important in terms of increasing the quality of life of patients and providing evidence for nursing practices by using it as a new method that can be applied in the care of cancer patients with chemotherapy-induced peripheral neuropathy. The aim of this research was to determine the effect of hand-foot exercises on the severity of pain, falls and quality of life associated with platinum-based therapy-related peripheral neuropathy in patients with colorectal cancer.

DETAILED DESCRIPTION:
Aim of the study:This study was conducted to determine the effect of hand-foot exercises on platinum-based therapy-related peripheral neuropathy-related pain severity, falls and quality of life in patients with colorectal cancer.

Design of the study:The research is a randomized controlled experimental study conducted to determine the effect of hand-foot exercises on platinum-based therapy-related peripheral neuropathy-related pain severity, falls and quality of life in patients with colorectal cancer.

Study place and date:The research was carried out in Gülhane Training and Research Hospital Medical Oncology Outpatient Chemotherapy Unit. Research data were collected between 25 April and 31 December 2022.

Sample and setting:The population of the study consists of patients diagnosed with colorectal cancer who received platinum-based treatment in Gülhane Training and Research Hospital Medical Oncology Outpatient Chemotherapy Unit between April 25 and December 31, 2022. The sample of the study consists of patients who were diagnosed with colorectal cancer in Gülhane Training and Research Hospital Medical Oncology Outpatient Chemotherapy Unit between April 25 and December 31, 2022, received at least 2 and maximum 7 cycles of platinum-based chemotherapy and accepted to participate in the study.

Measuraments:Research data were collected with Sociodemographic and Clinical Characteristics Form, Exercise Follow-up Form, EORTC QLQ-C30 scale, EORTC QLQ-CR29 scale, Chemotherapy-Induced Peripheral Neuropathy Assessment Tool, Numerical Pain Rating Scale, Fall Status Follow-up Form.

Ethical considerations:Ethics committee approval was obtained from Ankara University Ethics Committee for the conduct of the study. Institutional permission was obtained from Gülhane Training and Research Hospital, the institution where the research was conducted.Verbal and written informed consent was obtained from the patients who agreed to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older.
* Not having any physical or mental health problems that will prevent communication.
* Being conscious and cooperative.
* Being diagnosed with colorectal cancer.
* Receiving 2, 3, 4, 5, 6 or 7 cycles of platinum-based chemotherapy.
* Being treated with the FOLFOX regimen.
* Having chemotherapy-induced peripheral neuropathy according to CIPNAT (Chemotherapy-Induced Peripheral Neuropathy Assessment Tool). (Answering "yes" to the first 4 questions)
* Agree to participate in the research.

Exclusion Criteria:

* Receiving less than 2 cycles of platinum-based therapy.
* To be receiving platinum-based treatment at 8th cycle and above.
* Being diagnosed with a chronic disease (diabetes) that can lead to peripheral neuropathy.
* Experiencing neuropathic symptoms due to cervical or lumbar hernia.
* Having a habit of using alcohol constantly.
* Being on medication that masks neuropathy signs or may develop neuropathy symptoms. (Opioid, beta blocker, anticonvulsant, tricyclic antidepressant etc.)
* Having previously received neurotoxic chemotherapy (such as taxane, vinca alkaloids, bortezomib).
* To have had major surgery in the last 1 month.
* Not having the physical and mental ability to complete the research.
* Refusing to participate in the research. Drop out Criteria
* Changing the chemotherapy protocol.
* Not being able to apply the Hand-Foot Exercises Program regularly.
* Indicate that they want to withdraw from the research while the research is in progress.
* Not being reached while the research is in progress.
* Losing life while research is in progress.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Chemotheraphy induced peripheral neuropaty related Pain Severity | 0. week (begining of the study) - 8. week (end of the study)
  Hand-foot exercise program effects on platiunum based chemotheraphy induced peripheral neuropathy related pain severtiy- Numeric Pain Rating Scale
Chemotheraphy induced peripheral neuropaty related Falls | 0. week (begining of the study) - 8. week (end of the study)
  Hand-foot exercise program effects on platiunum based chemotheraphy induced peripheral neuropathy related falls-Fall Follow-up Form
Colorectal cancer patient's Quality of Life | 0. week (begining of the study) - 8. week (end of the study)
  Hand-foot exercise program effects on quality of life of patients-EORTC QLQ-C30, EORTC QLQ-CR29 scales
Chemotherapy Induced Peripheral Neuropathy Symptoms Assessment | 0. week (begining of the study) - 8. week (end of the study)
  Hand-foot exercise program effects on chemotheraphy induced peripheral neuropathy symptoms- CIPNAT tool

CONTACTS AND LOCATIONS:
Locations (1):
- Gülhane Training and Resarch Hospital, Ankara, Ankara/Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
There is not a plan to make individual participant data (IPD) available to other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: Audiences of the research, pollsters, ethical committees and official authorities, researchers

REFERENCES:
- [Background] Carozzi VA, Canta A, Chiorazzi A. Chemotherapy-induced peripheral neuropathy: What do we know about mechanisms? Neurosci Lett. 2015 Jun 2;596:90-107. doi: 10.1016/j.neulet.2014.10.014. Epub 2014 Oct 22. PMID 25459280
- [Background] Seretny M, Currie GL, Sena ES, Ramnarine S, Grant R, MacLeod MR, Colvin LA, Fallon M. Incidence, prevalence, and predictors of chemotherapy-induced peripheral neuropathy: A systematic review and meta-analysis. Pain. 2014 Dec;155(12):2461-2470. doi: 10.1016/j.pain.2014.09.020. Epub 2014 Sep 23. PMID 25261162
- [Background] Tofthagen CS, McMillan SC, Kip KE. Development and psychometric evaluation of the chemotherapy-induced peripheral neuropathy assessment tool. Cancer Nurs. 2011 Jul-Aug;34(4):E10-20. doi: 10.1097/NCC.0b013e31820251de. PMID 21242773
- [Background] Korosteleva TA, Veresova OV. [Proliferative activity and cytotoxic effect of mouse lymphocytes during the growth of transplanted melanoma B-16]. Eksp Onkol. 1984;6(1):53-5. Russian. PMID 6499732
- [Background] Humphries SE, Peacock RE, Talmud PJ. The genetic determinants of plasma cholesterol and response to diet. Baillieres Clin Endocrinol Metab. 1995 Oct;9(4):797-823. doi: 10.1016/s0950-351x(95)80161-8. PMID 8593126
- [Background] Masini G, Gherardi C, Dianda R. [Hydrogen dilution curves in the diagnosis of right heart short circuits]. Boll Soc Ital Cardiol. 1970;15(4):318-20. No abstract available. Italian. PMID 4920214
- [Background] Kaley TJ, Deangelis LM. Therapy of chemotherapy-induced peripheral neuropathy. Br J Haematol. 2009 Apr;145(1):3-14. doi: 10.1111/j.1365-2141.2008.07558.x. Epub 2009 Jan 16. PMID 19170681
- [Background] Russell WE, McGowan JA, Bucher NL. Partial characterization of a hepatocyte growth factor from rat platelets. J Cell Physiol. 1984 May;119(2):183-92. doi: 10.1002/jcp.1041190207. PMID 6715416
- [Background] Zholkiver KI, Musabaeva LI, Balmukhanov SB. [The use of the method of critical points for planning telegammatherapy in cancer of the esophagus]. Med Radiol (Mosk). 1969 May;14(5):58-64. No abstract available. Russian. PMID 5386000
- [Background] Tofthagen C, McAllister RD, McMillan SC. Peripheral neuropathy in patients with colorectal cancer receiving oxaliplatin. Clin J Oncol Nurs. 2011 Apr;15(2):182-8. doi: 10.1188/11.CJON.182-188. PMID 21444285
- [Background] Bakitas MA. Background noise: the experience of chemotherapy-induced peripheral neuropathy. Nurs Res. 2007 Sep-Oct;56(5):323-31. doi: 10.1097/01.NNR.0000289503.22414.79. PMID 17846553
- [Background] Dhawan S, Andrews R, Kumar L, Wadhwa S, Shukla G. A Randomized Controlled Trial to Assess the Effectiveness of Muscle Strengthening and Balancing Exercises on Chemotherapy-Induced Peripheral Neuropathic Pain and Quality of Life Among Cancer Patients. Cancer Nurs. 2020 Jul/Aug;43(4):269-280. doi: 10.1097/NCC.0000000000000693. PMID 30888982
- [Background] Duregon F, Vendramin B, Bullo V, Gobbo S, Cugusi L, Di Blasio A, Neunhaeuserer D, Zaccaria M, Bergamin M, Ermolao A. Effects of exercise on cancer patients suffering chemotherapy-induced peripheral neuropathy undergoing treatment: A systematic review. Crit Rev Oncol Hematol. 2018 Jan;121:90-100. doi: 10.1016/j.critrevonc.2017.11.002. Epub 2017 Nov 7. PMID 29198853
- [Background] Win MMTM, Fukai K, Nyunt HH, Linn KZ. Hand and foot exercises for diabetic peripheral neuropathy: A randomized controlled trial. Nurs Health Sci. 2020 Jun;22(2):416-426. doi: 10.1111/nhs.12676. Epub 2019 Dec 26. PMID 31876991
- [Derived] Eroglu I, Kutluturkan S. The effect of hand-foot exercises on chemotherapy-induced peripheral neuropathy-related pain, falls, and quality of life in colorectal cancer: A randomized controlled trial. Eur J Oncol Nurs. 2024 Aug;71:102641. doi: 10.1016/j.ejon.2024.102641. Epub 2024 Jun 15. PMID 38897103